CLINICAL TRIAL: NCT01341236
Title: Evaluation of Splanchnic Oximetry,Doppler Flow Velocimetry in the Superior Mesenteric Artery and Feeding Tolerance in VERY LOW BIRTH WEIGHT IUGR and NON-IUGR Infants Receiving Bolus Versus Continuous Enteral Nutrition
Brief Title: Near Infrared Spectroscopy (NIRS) and Superior Mesenteric Artery (SMA) Doppler Patterns as Predictor of Feeding Tolerance in Very Low Birth Weight (VLBW) IntraUterine Growth Restricted (IUGR) and NON IUGR Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Responsible Party: Principal Investigator, Valentina Bozzetti, Dr., San Gerardo Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Feeding VLBW
Record Dates: First submitted 2011-04-12; First posted 2011-04-25 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Infant, Very Low Birth Weight; Infant Malnutrition; Feeding Disorder of Infancy or Early Childhood; Splanchnic Oximetry; Splanchnic Oxygenation
Keywords: VLBW; IUGR; NIRS; enteral nutrition; superior mesenteric artery doppler
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous nutrition (Active Comparator)
  Interventions: Other: different nutrional regimen
- bolus nutrition (Active Comparator)
  Interventions: Other: comparison of different feeding regimens

INTERVENTIONS:
Other: different nutrional regimen — compare bolus versus intermittent nutrition
  Arms: continuous nutrition
Other: comparison of different feeding regimens — compare intermittent versus bolus nutrition
  Arms: bolus nutrition

SUMMARY:
This study aims at recruiting about twenty very low birth weight infants, either intrauterine growth restricted (IUGR) or NON-IUGR

STRATIFICATION:Population will be stratified in two groups: IUGR infants (approximately 10 children) and NON-IUGR infants (approximately 10 children).

PRIMARY ENDPOINT:To evaluate the changes in the intestinal perfusion determined by feeding in VLBW infants fed by 3 hours nasogastric nutrition (CN) or by bolus (BN).

SECONDARY ENDPOINT:

* To compare if changes in the intestinal perfusion induced by feeding are different between IUGR and NON-IUGR infants;
* To compare growth and nutritional status of the 2 groups by randomized arm.
* To evaluate if changes of intestinal perfusion and oximetry induced by feeding are related to baseline (< 72 hours of life) values of Doppler flow velocimetry and of Near Infrared Spectroscopy (NIRS). After birth, in the first 24 hours of life, and in the transitional period, between the 48th and 72nd hours of life, all infants' intestinal perfusion will be evaluated with NIRS and a doppler of the superior mesenteric artery will be executed.
* To test if changes in intestinal oximetry and perfusion can be reliable predictors of feeding intolerance (need of interruption of enteral feeding).

DESIGN: This is a randomized, non-pharmacological, single-center, cross-over study including 20 VLBW babies. Duration of the study: 24 months.

INCLUSION CRITERIA

* Weight at birth ranging: 700 - 1501 grams;
* Gestational age up to 25 weeks and 6 days;
* Written informed consent from parents or guardians

EXCLUSION CRITERIA

* Major congenital abnormality (severe heart or cerebral disease, chromosomopathies, severe renal malformations, any malformation or disease of the gastroenteric tract)
* Significant multi-organ failure prior to trial entry (perinatal asphyxia with renal, cardiac or cerebral impairment, DIC)
* Pre-existing cutaneous disease not allowing the placement of the probe

ELIGIBILITY:
Inclusion Criteria:

* Weight at birth ranging: 700 - 1501 grams;
* Gestational age up to 25 weeks and 6 days;
* Written informed consent from parents or guardians.

Exclusion Criteria:

* Major congenital abnormality (severe heart or cerebral disease, chromosomopathies, severe renal malformations, any malformation or disease of the gastroenteric tract)
* Significant multi-organ failure prior to trial entry (perinatal asphyxia with renal, cardiac or cerebral impairment, DIC)
* Pre-existing cutaneous disease not allowing the placement of the probe

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
changes in the intestinal perfusion determined by feeding in VLBW infants fed by 3 hours nasogastric nutrition (CN) or by bolus (BN). | 3 hours
  Evaluation of oximetry with splanchnic NIRS (difference of CSOR values and of rSO2s values) and perfusion with doppler of superior mesenteric artery (differences of peak sistolic and end-diastolic velocity, mean velocity, and pulsatility index) before, during ad after feeding.

SECONDARY OUTCOMES:
To compare of changes in the intestinal perfusion induced by feeding are different between IUGR and NON-IUGR infants; | 2 weeks; it's an average;it depends on the time necessary to achieve an enteral intake of 100 mL/Kg/die
  • To compare if changes in the intestinal perfusion induced by feeding are different between IUGR and NON-IUGR infants with NIRS (difference of CSOR values and of rSO2s values) and doppler of the superior mesenteric artery measurements (difference of peak sistolic and end-diastolic velocity, mean velocity, and pulsatility index) ;
• To compare growth and nutritional status of the 2 groups by randomized arm. | 2 months; it's an average;it depends on the time necessary to achieve the full enteral feeding and the 36th weeks of postconceptional age
  Measurements of body weight (grams), length and head circumference (cm) will be performed at predefined times: at birth, at the beginning of MEF, on the randomization day, at the achievement of full enteral feeding, at 28 days of life and at 36 weeks of gestational age
• To evaluate if changes of intestinal perfusion and oximetry induced by feeding are related to baseline (< 72 hours of life) values of Doppler flow velocimetry and of NIRS. | 2 weeks
  Comparison of the values of Doppler flow velocimetry of the superior mesenteric artery and of abdominal NIRS during feeding with those registered after birth, in the first 24 hours of life, and in the transitional period.
• To test if changes in intestinal oximetry and perfusion can be reliable predictors of feeding intolerance | 1 month; it's an average;it depends on the time necessary to achieve the full enteral feeding
  Time necessary to achieve full enteral feeding will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Paolo E Tagliabue, MD, Study Director — San Gerardo Hospital
Locations (1):
- NICU San Gerardo Hospital, Monza, MonzaBrianza, Italy

REFERENCES:
- [Derived] Bozzetti V, Paterlini G, De Lorenzo P, Gazzolo D, Valsecchi MG, Tagliabue PE. Impact of Continuous vs Bolus Feeding on Splanchnic Perfusion in Very Low Birth Weight Infants: A Randomized Trial. J Pediatr. 2016 Sep;176:86-92.e2. doi: 10.1016/j.jpeds.2016.05.031. Epub 2016 Jun 20. PMID 27339251
- [Derived] Bozzetti V, Paterlini G, Meroni V, DeLorenzo P, Gazzolo D, Van Bel F, Visser GH, Valsecchi M, Tagliabue PE. Evaluation of splanchnic oximetry, Doppler flow velocimetry in the superior mesenteric artery and feeding tolerance in very low birth weight IUGR and non-IUGR infants receiving bolus versus continuous enteral nutrition. BMC Pediatr. 2012 Jul 24;12:106. doi: 10.1186/1471-2431-12-106. PMID 22828032